CLINICAL TRIAL: NCT04126382
Title: The Efficacy of LISA Technology With Noninvasive Ventilation in the Treatment of Respiratory Distress Syndrome in Preterm Neonates
Brief Title: LISA vs INSURE in the Treatment of Respiratory Distress Syndrome in Preterm Infants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: The First Affiliated Hospital of University of Science and Technology of China (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Second Affiliated Hospital of Bengbu Medical College (Other); Fuyang people's hospital (Other); lixin people's hospital (Unknown); The Third People's Hospital of Bengbu (Other Government); Huaibei coal general hospital (Unknown); Bozhou people's hospital (Unknown); Luan people's hospital (Unknown); Huaibei maternal and child health hospital (Unknown); Huainan maternal and child health hospital (Unknown); Chizhou people's hospital (Unknown); Xuancheng people's hospital (Unknown); First Affiliated Hospital of Wannan Medical College (Other); Tongling People's Hospital (Other Government); Maanshan maternity and child care (Unknown); Wuhu first people's hospital (Unknown); Anqing Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LISA2020
Record Dates: First submitted 2019-10-04; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Preterm Infants
Keywords: NRDS; preterm infants; LISA; INSURE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INSURE (Active Comparator): Intubate-Surfactant-Extubate(INSURE) technique is a Important treatment in premature infants with RDS.
  Interventions: Procedure: Intubate-Surfactant-Extubate(INSURE)
- LISA (Experimental): Less invasive surfactant administration(LISA) technique is a Important treatment in premature infants with RDS.
  Interventions: Procedure: less invasive surfactant administration(LISA)

INTERVENTIONS:
Procedure: Intubate-Surfactant-Extubate(INSURE) — Infants are given an endotracheal intubation, with manual lung inflation in order to keep the oxygen supply，and the surfactant(kelisu,China Resources Shuanghe Pharmaceutical) was slowly instilled into the airway through the tracheal tube, and the tracheal tube was removed for non-invasive NCPAP(nasal continuous positive airway pressure)-assisted breathing.
  Arms: INSURE
Procedure: less invasive surfactant administration(LISA) — Infants are spontaneously breathing with nasal CPAP(continuous positive airway pressure) support without manual lung inflation and surfactant(kelisu,China Resources Shuanghe Pharmaceutical) is administered through vocal cords via a smaller catheter.
  Arms: LISA

SUMMARY:
To evaluate the efficacy of less invasive surfactant administration（LISA ）technique in the treatment of neonatal respiratory distress syndrome（NRDS） by comparing with the traditional Intubate-Surfactant-Extubate（INSURE） technique.

DETAILED DESCRIPTION:
Background: Neonatal Respiratory distress syndrome (NRDS) is the most common cause of respiratory problems in premature babies. Surfactant administration involved with endotracheal intubation and mechanical ventilation has proven to be a effective treatment, however, it is associated with a risk of barotrauma, volutrauma and bronchopulmonary dysplasia(BPD). In recent years, some studies have demonstrated that prophylactic INSURE did not lead to a higher survival without BPD, and LISA technique is recommended. However there is no multicenter and Large sample research about it. The aim of this multicenter trial is to compare the efficacy between LISA-treated and INSURE-treated premature Preterm babies with respiratory distress syndrome(RDS).

Methods/Design：In this multicenter, randomized, cohort, prospective trial, 200 preterm infants from 18 neonatal intensive care units in AnHui province whose gestational age (GA) less than 32 weeks with a diagnosis of RDS will be randomized to LISA-treated group and INSURE-treated group.

The primary outcomes include rate of intubation,incidence of bronchopulmonary dysplasia(BPD).The secondary outcomes include arterial blood gas analysis,severity of RDS,the incidence of Patent ductus arteriosus(PDA),Pneumothorax,Abdominal Distention,Neonatal Necrotizing Enterocolitis(NEC,>Stage II), Retinopathy of Prematurity( ROP,≥ Stage II), Intraventricular Hemorrhage (IVH, ≥ Grade Ⅲ), Periventricular Leukomalacia(PVL) , mortality, days on noninvasive respiratory support,days on supplemental oxygen and days of hospitalization.Other secondary outcomes include scores of Gesell development Scales of infant development at 3 years of corrected age.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) less than 32 weeks
* diagnosis of RDS. The diagnosis of RDS will be based on clinical manifestations (Progressive dyspnea, nasal flaring and or grunting), chest X-ray findings and need for noninvasive ventilation support(fraction of inspired oxygen>40％) in 6 hours after birth
* informed parental consent has been obtained

Exclusion Criteria:

* severe RDS have been treated with endotracheal intubation,surfactant and mechanical ventilation
* major congenital malformations or complex congenital heart disease
* Pulmonary hemorrhage
* Cardiopulmonary failure
* septicemia, Intraventricular Hemorrhage (IVH, ≥ Grade Ⅲ), and Congenital genetic metabolic disease
* transferred out of the NICUs(neonatal intensive care units) with surgical treatment or other intervention

Ages: 25 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of intubation | during the first 3 days after birth
  The criteria for endotracheal mechanical ventilation were as follows: severe apnea and bradycardia (defined as recurrent apnea with > 3 episodes per hour associated with heart rate < 100/min, a single episode of apnea that required bag and mask ventilation), hypoxia (FiO2>0.6 with PaO2<50mmHg or TcSO<0.85), severe respiratory acidosis (PaCO2 > 60 mmHg with pH<7.20).
The incidence of bronchopulmonary dysplasia | at a post-menstrual age of 36 weeks or at discharge
  BPD was diagnosed and classified based on the Practical neonatology 4th edition:Need for O2 supplementation(FiO2>0.21) for at least 28 days after birth.

SECONDARY OUTCOMES:
Effect on of arterial blood gas analysis | during the whole procedure of surfactant replacement,up to 3 days after birth
  The improvement of PaO2 and PaCO2 in two groups children with LISA technique
The Incidence of Patent ductus arteriosus | during hospitalization, up to 60 days
  PDA was diagnosed based on echocardiography
The Incidence of Pneumothorax | during non-invasive ventilation, up to 30 days
  Pneumothorax was diagnosed based on clinical manifestations and features of chest x-ray
The Incidence of Abdominal Distention | during non-invasive ventilation, up to 30 days
  Abdominal circumference was measured 3 times a day during non-invasive ventilation
The Incidence of Neonatal Necrotizing Enterocolitis(>Stage II) | during hospitalization, up to 60 days
  Neonatal Necrotizing Enterocolitis was diagnosed by clinical manifestations and features of abdominal x-Ray based on the Practical neonatology 4th edition
The Incidence of Retinopathy of Prematurity( ≥ Stage II) | at a post-menstrual age of 36 weeks or at discharge
  The criteria for Retinopathy of prematurity (>Stage II); extraretinal fibrovascular proliferation neovascularization extends from ridge into the vitreous.
The Incidence of Intraventricular Hemorrhage (IVH, ≥ Grade Ⅲ) | during hospitalization, up to 60 days
  The criteria for intraventricular hemorrhage (IVH, ≥ grade Ⅲ): intraventricular hemorrhage with ventricular dilatation and intraventricular hemorrhage with paren-ehymal hemorrhage.
The Incidence of Periventricular Leukomalacia | during hospitalization, up to 36 months
  Periventricular Leukomalacia was diagnosed based on cranial MRI
Predischarge Mortality | during hospitalization, up to 60 days
The Time of Non-invasive Ventilation | during hospitalization, up to 60 days
  Hours
Days on supplemental oxygen | during hospitalization, up to 60 days
  Days
Length of Hospitalization | during hospitalization, up to 60 days
  Days

CONTACTS AND LOCATIONS:
Overall Officials: Pan jiahua, PhD, Study Director — Director of pediatric department of the First Affiliated Hospital of University of Science and Technology of China

IPD SHARING:
Plan to Share IPD: Undecided